CLINICAL TRIAL: NCT07363889
Title: Vitrectomy Machine Versus Spring Loaded Syringe for Active Silicon Oil Extraxtion
Brief Title: Spring Loaded Syringe for Active Silicon Oil Extraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Abdalsadek Ahmed Sinjab, Lecturer of Ophthalmology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-25-11-9PD
Record Dates: First submitted 2025-12-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Retinal Detachment
Keywords: Pars plana vitrectomy; Silicon oil tamponade; Silicon oil extraction
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Conventional technique using vitrectomy machine
  Interventions: Device: Vitrectomy machine
- Group B (Active Comparator): Spring loaded syringe for silicon oil extraction
  Interventions: Device: Spring loaded syringe

INTERVENTIONS:
Device: Vitrectomy machine — Active silicon oil extraction through 23G pars plana system vitrectomy machine
  Arms: Group A
Device: Spring loaded syringe — 5 mml syringe with spring in its plunger and rubber connection
  Arms: Group B

SUMMARY:
The aim of our study is to compare between two techniques used for active SOR. The outcomes include efficiency and safety.

Patients with silicon filled eyes and prepared for SOR 540 eyes of 505 patients (one eye in 470 patients, and both eyes in 35 patients) were enrolled in the study.

All eyes underwent SOR using 23-Gauge PPV. The eyes were classified according to the surgical technique used for SOR into two groups:- Group A: SOR was performed using SO extraction program built in Optikon vitrectomy device Group B: SOR was performed using modified spring loaded syringe.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected previously to pars plana vitrectomy with silicon oil tamponade.

Exclusion Criteria:

* Recurrent retinal detachment
* Previous scleral buckling
* Previous glaucoma surgery
* Bleeding tendencies
* Anterior staphyloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | During the surgical procedure and up to 3 months postoperative
  Incidence of operative and postoperative complications in both groups

OTHER OUTCOMES:
Time required for silicon oil extraction | From beginning of silicon oil extraction until complete extraction, It is recorded for every individual surgical procedure
  Total time in seconds needed to completely remove silicon oil, it is recorded by an assistant.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All unidentified IPD will be available and can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year, and will be available for unlimited time.
Access Criteria: All researchers will be able to access IPD through trial registry website or via r quest through our individual emails.